CLINICAL TRIAL: NCT04778735
Title: Investigation of Mortality, Morbidity and Risk Factors After Pediatric Liver Transplantation: A Retrospective Study
Brief Title: Investigation of Mortality, Morbidity and Risk Factors After Pediatric Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Bahçelievler Hospital (Other)
Responsible Party: Principal Investigator, Kamil Yalçın Polat, Prof.Dr., Memorial Bahçelievler Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MemorialBahcelievler
Record Dates: First submitted 2021-02-24; First posted 2021-03-03 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-02

CONDITIONS: Liver Transplantation; Liver Diseases; Biliary Atresia; Morbidity;Infant; Mortality
MeSH Terms: conditions — Liver Diseases; Biliary Atresia | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric Patients with Liver Transplantation (Other)
  Interventions: Procedure: Liver Transplantation

INTERVENTIONS:
Procedure: Liver Transplantation — Liver Transplantation is performed under spesific conditions to increase the life time of patients with liver diseases.

SUMMARY:
The Department of Organ Transplantation in Memorial Hospitals has started Pediatric Liver Transplantation Program in 2016. As of the end of 2020, we have performed 169 pediatric liver transplantation. The aim of this study is to investigate the overall mortality, morbidity and risk factors for adverse outcomes in pediatric liver transplantation. The patients' records will be retrospectively scanned and the data will be gathered.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with liver transplantation (<18 years)

Exclusion Criteria:

* Patients with incomplete medical records will be excluded

Ages: 0 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 207 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Survival | 1 minutes
  Patient and graft survival ratios

SECONDARY OUTCOMES:
Perioperative informations | 5 minutes
  Perioperative informations such as blood loss and blood transfusion
Blood Tests | 15 minutes
  Blood markers that evaluated at the pre and post operative phase such as Internation Normalized Ratio (INR), total bilirubin and albumin values.
Postoperative Complications | 5 minutes
  Postoperative Complications such as sepsis or hepatic artery thrombosis
Postoperative informations | 10 minutes
  Postoperative informations such as initial hospital stay, ICU stay or mechanic ventilation time

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Bahçelievler Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No